CLINICAL TRIAL: NCT04924959
Title: Construction and Validation of Risk Prediction Model for PICC Catheter Displacement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-205
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cancer Patients With PICC

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling Group
  Interventions: Other: Logistic Regression Analysis
- Validation Group

INTERVENTIONS:
Other: Logistic Regression Analysis — Using logistic regression analysis to analyze the independent risk factors of PICC catheter displacement
  Groups: Modeling Group

SUMMARY:
The occurrence of PICC catheter displacement is caused by many factors. In order to predict the risk of PICC and early warn high-risk patients, this study prospectively included patients with PICC catheter in a three Grade-A hospitals in June 2019, analyzed a variety of related factors, built a scientific and effective risk prediction model of PICC catheter displacement, and verified the goodness of fit and differential validity of the model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PICC

Exclusion Criteria:

* Patients with primary ectopia during PICC catheterization
* Patients with secondary ectopic adjusting length of catheter exposure
* Patients with mental illness and cognitive impairment
* Patients with incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with PICC
Sampling Method: Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Prediction Model of PICC catheter displacement | 3 years
  A mathematical model for predicting PICC catheter displacement

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affilicated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China